CLINICAL TRIAL: NCT00902941
Title: Reversibility of Olfactory Loss in Patients With Idiopathic Parkinson's Disease Following Treatment With Rasagiline
Brief Title: Olfaction in Patients With Parkinson's Disease Following Treatment With Rasagiline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUD-Olfact-035; 2008-005085-30
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s disease; olfaction; rasagiline; smell testing
MeSH Terms: conditions — Parkinson Disease; Anosmia | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Experimental)
  Interventions: Drug: Azilect 1mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilect 1mg — 1 mg daily orally for 120 days
  Arms: Rasagiline
Drug: Placebo — 1 mg daily orally for 120 days
  Arms: Placebo

SUMMARY:
There is convincing evidence from numerous studies using both psychophysical and electrophysiological approaches that olfaction is markedly reduced in Parkinson´s disease (PD). Data on the prevalence of olfactory dysfunction in PD however, range from 45% and 49% in the pioneering studies of Ansari & Johnson, and Ward, respectively, up to 74% in the work of Hawkes et al., or as high as 90% in a study published by Doty et al. Quality of life, safety, and interpersonal relations, as well as food behavior/nutritional intake are severely altered in a large proportion of patients with olfactory loss. Thus, the same can be assumed in patients with Parkinson's disease. If it was possible to improve olfactory function this would appear as a significant effect in patients with Parkinson's disease. Provided the study would reveal an improvement of olfactory function following therapy with rasagiline, this would have tremendous worldwide impact on the use of this drug. Considering the frequency of PD a very large number of patients would benefit from these findings, especially in terms of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson´s disease, Hoehn & Yahr stage ≤ III
* aged 18-64 yrs
* hyposmia/functional anosmia defined as TDI<30
* written consent

Exclusion Criteria:

* congenital olfactory loss
* significant infections of the nose and nasal sinuses
* diseases/states apart from PD which may significantly affect olfactory function, e.g., asthma, head trauma etc.
* dementia, psychiatric illness, addictive behaviour
* smoker
* severe liver disease
* pregnant or breastfeeding women
* any contraindication for the treatment with Rasagiline
* women without reliable contraception

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2009-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
olfactory function | 4 months

SECONDARY OUTCOMES:
quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Reichmann, MD, PhD, Principal Investigator — University of Dresden Medical School
Locations (1):
- University of Dresden Medical School, Smell & Taste Centre, Dept. of Neurology, Dresden, Germany